CLINICAL TRIAL: NCT01830049
Title: Differential Plasma MicroRNA Profiles in ED and Normal Erectile Function in Older Males
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Nanjing Medical University (Other)
Responsible Party: Principal Investigator, Feng Pan, MD., Nanjing Medical University
Other Study IDs: NJU2013024; 2013024 (Other: Nanjing University, Medical School)
Record Dates: First submitted 2013-04-09; First posted 2013-04-11 (Estimated); Last update posted 2013-04-11 (Estimated); Status verified 2013-04

CONDITIONS: Erectile Dysfunction
MeSH Terms: conditions — Erectile Dysfunction

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional

GROUPS / COHORTS (3):
- Group I: Older males with ED
  Interventions: Other: Take blood
- Group II: Older males with normal erectile function
  Interventions: Other: Take blood
- Gourp III: Young males with normal rectile function
  Interventions: Other: Take blood

INTERVENTIONS:
Other: Take blood

SUMMARY:
Erectile dysfunction (ED) is strongly associated with aging. With the rapidly expanding aging population and the increase in life expectancy, an increase in the prevalence of ED is expected in the years to come. Currently, the mechanism of ED is not fully understood. MicroRNAs (MiRNA) are endogenous small RNA molecules that control gene expression post-transcriptionally. It has been included in many in vitro physiology and pathophysiology processes, which also involved in the process of ED. This research was designed to investigate the differential plasma MiRNA profiles in ED and normal erectile function in older males. The results might tell us which MiRNA and how did it involved in the process of ED in aging.

ELIGIBILITY:
Inclusion Criteria:

* older males with erectile dysfunction

Exclusion Criteria:

* have some other general diseases, e.g. hypertension, vascular diseases, depression, chronic kidney disease, diabetes.

Ages: 20 Years to 80 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Group I: older males came to our clinic for diagnosis and treatment of ED. Group II: older males came to our clinic for physical examination and the erectile function was normal.
  Group III: young males came to our clinic for physical examination and the erectile function was normal.
Sampling Method: Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2013-03; Primary Completion 2013-07 (Estimated); Study Completion 2013-08 (Estimated)

PRIMARY OUTCOMES:
Gene chips | 30 days

SECONDARY OUTCOMES:
RT-PCR | 15 days

CONTACTS AND LOCATIONS:
Locations (1):
- Nanjing Gulou Hospital affiliated to Nanjing University, Medical School, Nanjing, Jiangsu, China